CLINICAL TRIAL: NCT03195933
Title: Learning, Neural Signaling of Cortisol, and Early Adversity in Depression
Brief Title: Depression, Adversity, and Stress Hormones (DASH) Study
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-0897; R01MH094478 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Depression
Keywords: Depression; Childhood Adversity; Childhood Abuse; Cortisol; Emotional Memory; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Depression | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cortisol first, Placebo second (Experimental): Single oral administration of 20 mg cortisol capsule to pharmacologically elevate cortisol levels during first functional magnetic resonance imaging (fMRI) session; Identically appearing placebo capsule during second fMRI session.
  Interventions: Other: Cortisol; Other: Placebo
- Placebo first, Cortisol second (Experimental): Placebo capsule during first fMRI session; Single oral administration of 20 mg cortisol capsule to pharmacologically elevate cortisol levels during second fMRI session.
  Interventions: Other: Cortisol; Other: Placebo

INTERVENTIONS:
Other: Cortisol — We compared placebo vs. 20 mg oral dose of cortisol, which pharmacologically elevated cortisol levels.
Other: Placebo — We compared placebo vs. 20 mg oral dose of cortisol, which pharmacologically elevated cortisol levels.

SUMMARY:
The stress-related hormone cortisol has been studied in depression for decades. However, relatively little is known about the role of cortisol in psychological features of depression. Basic research shows that cortisol modulates brain processes that are highly relevant to depression (especially the neural substrates of negative biases in learning and memory formation). However, very few studies have directly examined the effects of cortisol on neural circuitry of learning in depressed humans. In addition, the effects of cortisol on the neural substrates of learning differ for males and females. The toll of depression is especially high in women, who are roughly twice as likely as men to suffer from depression. Thus, the primary goal of this project is to investigate the effects of cortisol on the neural circuitry of learning in depressed women.

A secondary goal is to investigate whether early life adversity moderates cortisol's effects on the neural circuitry of learning. Animal data suggests that early life adversity causes life-long biases toward learning in threatening conditions associated with elevated cortisol. In addition, new data from humans suggests that alterations in cortisol traditionally ascribed to depression may stem in part from early adversity rather than depression per se. Thus, this study will examine effects of cortisol on the neural circuitry of learning in depressed and healthy women with and without history of early life adversity.

The study will use pharmacological manipulation of cortisol levels (compared to placebo) during measurement of brain activity at rest and during memory encoding of emotional and neutral stimuli. The study will also measure whether cortisol alters the negative biases in emotional memory often seen in depression. In doing so, the study will examine the role of cortisol in neural networks associated with emotional learning that are often implicated in depression.

Medications that target cortisol receptors in the brain may be beneficial in the treatment of depression. However, this knowledge has yet to inform clinical practice, and mechanisms of action of these medications are not well understood. This project is significant because it provides the prerequisite knowledge (and develops a paradigm) that can be used in the future in the development of more effective targeted intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 to 45 years of age
* English fluency
* Able to lie still on their back for up to 90 minutes
* Willing and able to return for all visits
* Able to provide written informed consent prior to participation
* In good physical health as determined on basis of medical history
* If a nicotine user, able to refrain from nicotine use for 2 hours prior to fMRI scanning and throughout the scan visits
* Additional criteria for never-depressed participants: Free of current or past Diagnostic and Statistical Manual (DSM) IV diagnoses of Major Depressive Disorder (MDD), Dysthymia, or other Depressive Disorder. Never-depressed participants may have past or current psychopathology other than depressive disorders that does not cause significant impairment in functioning and that would not interfere with study participation, be exacerbated by study participation, or introduce scientific difficulties, for example, history of complicated bereavement or history of time-limited alcohol abuse that does not represent a lasting substance use disorder
* Additional criteria for participants with MDD: Meet DSM-IV criteria for MDD (single or recurrent) as determined by a Structured Clinical Interview for DSM-IV (SCID)
* Additional criteria for depression-prone participants: Does not meet criteria for current MDD, but meets at least one of the following requirements:

  1. Meets DSM-IV criteria for past MDD (single or recurrent) as determined by a SCID interview
  2. Meets DSM-IV criteria for Depressive Disorder Not Otherwise Specified (NOS)
  3. Meets DSM-IV criteria for Dysthymia
  4. Has a Beck Depression Inventory (BDI) score of 14 or higher

Exclusion Criteria:

* Current use of any anti-depressant or psychotropic medication while participating in Visits 1-6 and Home Saliva Collection; treatment with electroconvulsive therapy (ECT) within the past 3 months; use of any anti-depressant within 14 days of participation, fluoxetine within 30 days of participation, or any other psychotropic drug within a timeframe based on the half-life of the particular drug
* Using hormonal contraceptives while participating in Visits 1-6 and Home Saliva Collection
* Using any medication that affects central nervous system (CNS) function for 2-4 weeks prior to testing and during participation in Visits 1-6 and Home Saliva Collection
* Using any illicit drug for 4 weeks prior to testing and during participation in Visits 1-6 and Home Saliva Collection
* Using any steroid, anti-histamine, nasal spray (which includes corticosteroids), or topical hydrocortisone cream/gel that affects the hypothalamic-pituitary-adrenal (HPA) axis for 2-4 weeks prior to testing and throughout the duration of the study
* History of seizures, diabetes, hypertension, neurological problems, and/or cardiac problems
* Metallic implants (i.e., prostheses, shrapnel, or aneurysm clips) or electronic implants (i.e., cardiac pacemakers) that are contraindicated for MRI
* Any clinically significant abnormalities on medical history or physical exam
* Currently pregnant, trying to become pregnant, breastfeeding, within a six-month window following pregnancy or breastfeeding, sexually active without an acceptable method of birth control (e.g., abstinence, male vasectomy, female sterilization, condom)
* Post-menopausal and peri-menopausal women
* Women with highly irregular menstrual cycles (e.g., more than 60 days between periods or less than 14 days between periods)
* Individuals who work the "night shift" (e.g., between the hours of 11 pm and 7 am) will be excluded due to potential variability in cortisol levels determined by sleep schedule
* Heavy nicotine user (e.g., smokes more than a pack/day)
* Unable to fit comfortably in the MRI simulator and/or scanner (e.g., BMI greater than approx. 38)
* Weight greater than approx. 250 lbs
* Lifetime history of mania or psychosis
* At risk for suicide as determined by a clinical interview
* Gross impairment in functioning
* Claustrophobia
* Frank Axis I or Axis II psychopathology that would interfere with study participation, become exacerbated by study participation, or introduce scientific difficulties

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Emotional Memory after Cortisol Administration | 15 minute memory assessment that takes place 2 days after cortisol administration MRI scan visit
  Memory for emotional pictures encoded during the cortisol administration MRI scan

SECONDARY OUTCOMES:
Neural Function | 90 minute scan session
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: Heather C. Abercrombie, Ph.D., Principal Investigator — University of Wisconsin School of Medicine & Public Health

IPD SHARING:
Plan to Share IPD: Yes
We will make our data publicly available on a password protected website after the data are collected and analyzed, and manuscripts presenting data testing our hypotheses are accepted for publication. These data will be thoroughly de-identified. Several classes of data will be made available, including self-report, behavioral, diagnostic, hormonal, and summary data from our physiological and imaging datasets.

REFERENCES:
- [Derived] Gaffey AE, Walsh EC, Ladd CO, Hoks RM, Abercrombie HC. Alterations in Systemic and Cognitive Glucocorticoid Sensitivity in Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Mar;4(3):310-320. doi: 10.1016/j.bpsc.2018.11.007. Epub 2018 Dec 4. PMID 30686583
- [Derived] Abercrombie HC, Frost CP, Walsh EC, Hoks RM, Cornejo MD, Sampe MC, Gaffey AE, Plante DT, Ladd CO, Birn RM. Neural Signaling of Cortisol, Childhood Emotional Abuse, and Depression-Related Memory Bias. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Mar;3(3):274-284. doi: 10.1016/j.bpsc.2017.11.005. Epub 2017 Nov 22. PMID 29486869